CLINICAL TRIAL: NCT03286933
Title: Yoga Therapy for Adolescents With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Adina, Adina Schwartz, MA, OTR/L, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-17-00037
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Adolescent Juvenile Idiopathic Arthritis; Yoga Therapy
Keywords: yoga therapy; JIA; quality of life; pain management
MeSH Terms: conditions — Agnosia | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga therapy intervention (Experimental): Participants will participate in weekly yoga therapy sessions and have the opportunity to use the home video online.
  Interventions: Behavioral: yoga

INTERVENTIONS:
Behavioral: yoga — 75 minute weekly group yoga classes for 8 weeks. Home program online.

SUMMARY:
The purpose of the study is to better understand the effects of a yoga program on adolescents with juvenile idiopathic arthritis (JIA). The investigators want to learn whether or not a yoga therapy based program will decrease pain and improve quality of life in patients with JIA.

This is an 8-week program with home program of online videos.

DETAILED DESCRIPTION:
This is an 8-week program consisting of weekly yoga therapy classes in a public studio. The classes are led by a pediatric occupational therapist who is also a certified internationally accredited yoga therapist (C-IAYT). The initial and final sessions will include an Rheumatologist MD evaluation including a physician global assessment and joint damage assessment (JADI) and visual assessment (VAS). A Visual Analog Pain Scale will and Peds Quality of Life Questionnaire-Arthritis Module 4.0 will be administered. Each yoga class is 75 minutes to include a set-sequence of postures including breathing exercises and final corpse pose (final relaxation).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with formal diagnosis of JIA, speak and understand English, can get on/off floor independently.

Exclusion Criteria:

* Dependent on assistive device for ambulation; does not understand English, does not have a diagnosis of JIA.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-06 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Peds QL-Arthritis Module 4.0 | 8 weeks
  Measures perceived quality of life for adolescents with arthritis
Visual Analog Pain Scale | 8 weeks
  Visual marker of perceived pain
Visual Assessment | 8 weeks
  Physician visual assessment
Joint Damage Assessment (JADI) | 8 weeks
  assessment of joints

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Participants will be coded and all data will be connected to their code. No names will be used after recruitment.